CLINICAL TRIAL: NCT02877641
Title: Effect of Once Daily Oral Vitamin D3 Supplementation on Inspiratory Muscle Strength in Vitamin D3-Deficient COPD Patients
Brief Title: Cholecalciferol Supplementation in Strengthening Inspiratory Muscles in Cholecalciferol-Deficient Patients With Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: I 240913; NCI-2016-00524 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 240913 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH); P50CA090440 (NIH)
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Muscle Weakness
Keywords: Current Smoker; Former Smoker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscle Weakness; Smoking Cessation | interventions — Cholecalciferol; Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (multivitamin, placebo) (Active Comparator): Patients receive a placebo and multivitamin orally each day for 52 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Dietary Supplement: Multivitamin; Other: Placebo; Other: Questionnaire Administration
- Supplementation arm (multivitamin, cholecalciferol) (Experimental): Patients receive a multivitamin and cholecalciferol supplement orally each day for 52 weeks.
  Interventions: Dietary Supplement: Cholecalciferol; Other: Laboratory Biomarker Analysis; Dietary Supplement: Multivitamin; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Given PO
  Other Names: 9,10-Secocholesta-5,7,10(19)-trien-3-ol; Calciol; Delsterol; Vitamin D3
  Arms: Supplementation arm (multivitamin, cholecalciferol)
Other: Laboratory Biomarker Analysis — Correlative studies
Dietary Supplement: Multivitamin — Given PO
  Other Names: Geritol; Vitamin Supplements (NOS)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Control arm (multivitamin, placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase IIb randomized trial studies how well cholecalciferol (vitamin D3) supplementation works in strengthening inspiratory muscles in cholecalciferol-deficient patients with chronic obstructive pulmonary disease (COPD). Cholecalciferol supplementation may help reduce the risk of developing lung cancer and strengthen the diaphragm in cholecalciferol-deficient patients with COPD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the effect of D vitamin (vitamin D3) supplementation on inspiratory muscle strength in vitamin D3-deficient chronic obstructive pulmonary disease (COPD) patients. (Roswell Park Cancer Institute [RPCI]/University at Buffalo [UB] study) II. To establish the 12 month conversion rate. (University of Pittsburgh Cancer Institute [UPCI] study)

SECONDARY OBJECTIVES:

I. To establish the effect of vitamin D3 supplementation on peripheral muscle strength and exercise capacity in vitamin D3-deficient COPD patients. (RPCI/UB study) II. To establish the 3 and 6-month conversion rates. (UPCI study) III. To examine whether vitamin D3 supplementation is equally effective in COPD patients who are current versus former smokers. (UPCI study)

TERTIARY OBJECTIVES:

I. To explore the effects of vitamin D3 supplementation in COPD patients on biomarkers of lung cancer risk, inflammation, and pulmonary function. (UPCI study)

OUTLINE: Patients are randomized to 1 of 2 arms.

CONTROL ARM: Patients receive a placebo and multivitamin orally (PO) once daily (QD) for 52 weeks.

SUPPLEMENTATION ARM: Patients receive a multivitamin and cholecalciferol supplement PO QD for 52 weeks.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Current or ex-smoker with at least a 10-year pack history
* COPD, defined as forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) < 70% and FEV1% predicted < 80%
* 25-hydroxy vitamin D3 (25[OH]D3) level less than 20 ng/mL prior to study initiation
* Willingness to comply with study guidelines
* Willingness to avoid alternative/additional vitamin D3 supplementation for the duration of the trial
* Subject must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Personal history of lung cancer or head and neck cancer
* History of malabsorption syndrome (e.g., pancreatic insufficiency, celiac disease, or tropical sprue)
* History of known thyroid disease
* History of known sarcoid disease
* History of known abnormalities in calcium metabolism
* Hypercalcemia (serum calcium in excess of laboratory upper limit normal [ULN])
* Self-reported consumption of more than 4 alcoholic drinks per day
* Use of anti-seizure medications phenobarbital or phenytoin, which can disrupt vitamin D metabolism
* History of known renal dysfunction
* History of known nephrolithiasis (kidney stones)
* Current use of supplemental oxygen
* Inability to exercise due to musculoskeletal issue, osteoarthritis or underlying cardiac disease
* Current participation in a cancer intervention prevention study, except for smoking cessation
* Any condition which in the Investigator's opinion deems the subject an unsuitable candidate to receive study drug
* Inability to swallow pills
* Vitamin D supplementation > 2,000 IU/day of vitamin D within 30 days prior to enrollment
* Positive Pregnancy Test

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-04-16 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Conversion rate, defined as the proportion of patients whose baseline cholecalciferol deficiency is corrected (UPCI study) | At 12 months
  75% will be considered a success.
Inspiratory muscle strength assessed by respiratory capacity (RPCI/UB study) | Baseline to 24 weeks
  Will be analyzed using linear mixed model by regressing the repeated outcome on the group indicator (treatment or control) and other appropriate covariates. Appropriate within-subject covariance will be determined from an exploratory study. The effect of vitamin D3 supplementation will be tested using an approximate t-test.

SECONDARY OUTCOMES:
Change in exercise capacity assessed by respiratory exercise tests (RPCI/UB study) | Baseline to 24 weeks
  Peak oxygen consumption will be used to establish cardiovascular fitness. Breath-by-breath measurements of minute ventilation, tidal volume, breathing frequency, end tidal carbon dioxide, carbon dioxide production and oxygen consumption will be continuously measured.
Change in peripheral muscle strength assessed by the elbow flexion test (RPCI/UB study) | Baseline to 24 weeks
  The elbow flexion test (upper extremity) requires participants to curl a standard 8 lb weight as many times as possible in a 30 second time period.
Conversion rate, defined as the proportion of patients whose baseline cholecalciferol deficiency is corrected (UPCI study) | At 3 months
  Efficacy in in COPD patients who are current versus former smokers will be compared.
Conversion rate, defined as the proportion of patients whose baseline cholecalciferol deficiency is corrected (UPCI study) | At 6 months
  Efficacy in in COPD patients who are current versus former smokers will be compared.
Change in peripheral muscle strength assessed by squat test (RPCI/UB study) | Baseline to 24 weeks
  This functional sit-to-stand test measures lower extremity strength. Participants will perform as many sit-to-stand repetitions from a standard height chair in 60 seconds as possible.

OTHER OUTCOMES:
Change in correlative biomarkers of lung cancer risk, inflammation, and pulmonary function (UPCI study) | Baseline to up to 1 year
  The vitamin D3 supplementation group will be compared to the placebo control group using two-sample t-tests at each time point for preliminary analysis. The correlation between muscle strength and the correlative biomarkers will be explored using Pearson correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Mahoney, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States